CLINICAL TRIAL: NCT00005715
Title: Community Intervention for Minority Children With Asthma
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4924; R01HL045312 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2000-05

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To test the effectiveness of school-based asthma education interventions, community-based asthma health workers' programs and the combination of these on asthmatic children. Also, to examine the separate and combined impact of asthma interventions designed to address problems associated with effective asthma self-management amd difficulties in establishing and maintaining continuity of medical care.

DETAILED DESCRIPTION:
BACKGROUND:

Asthma is a leading cause of childhood illness that disproportionately affects minority children. The causes of higher hospitalization and death rates among minority children with asthma are not understood. It is commonly assumed that barriers related to poverty underlie this public health issue. Two proposed causes of this increased morbidity and mortality are problems associated with effective asthma self-management and difficulties in establishing and maintaining continuity of medical care.

The study was part of a demonstration and education initiative "Interventions for Control of Asthma Among Black and Hispanic Children" which was released by the NHLBI in June 1989.

DESIGN NARRATIVE:

A school-based asthma self-management program was developed to promote children's self-management skills within predominately minority schools. A community-based asthma health worker program was developed to assist minority families in establishing and maintaining asthma health care within the community. It was hypothesized that the most effective control of asthma would be achieved with the combination of these two interventions. Twenty elementary schools each in inner-city Baltimore, Maryland and inner-city Washington D.C. served as study sites. Asthmatic children grades 1-5 were identified by school records and parent surveys. After obtaining consent, schools were randomly assigned to one of four intervention groups: 1) a control/minimal intervention, 2) a school-based asthma education program, 3) a community-based asthma health worker program, and 4) a combined intervention that included both the school-based education program and the community-based health worker program. The duration of both the school program and the Community health worker program was twelve months. Baseline measures were collected after obtaining consent and prior to school randomization. Followup measures were collected from children and families at 6, 12, 18, and 24 months. Data were collected on hospitalization, emergency or urgent care, acute episodes, health care utilization, medications, school absences, academic performance, self-esteem, self and family asthma management, and family coping.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-08; Study Completion 1995-07 (Actual)

REFERENCES:
- [Background] Butz AM, Malveaux FJ, Eggleston P, Thompson L, Schneider S, Weeks K, Huss K, Murigande C, Rand CS. Use of community health workers with inner-city children who have asthma. Clin Pediatr (Phila). 1994 Mar;33(3):135-41. doi: 10.1177/000992289403300302. PMID 8194287
- [Background] Huss K, Rand CS, Butz AM, Eggleston PA, Murigande C, Thompson LC, Schneider S, Weeks K, Malveaux FJ. Home environmental risk factors in urban minority asthmatic children. Ann Allergy. 1994 Feb;72(2):173-7. PMID 8109808
- [Background] Eggleston PA, Malveaux FJ, Butz AM, Huss K, Thompson L, Kolodner K, Rand CS. Medications used by children with asthma living in the inner city. Pediatrics. 1998 Mar;101(3 Pt 1):349-54. doi: 10.1542/peds.101.3.349. PMID 9480996
- [Background] Schneider SL, Richard M, Huss K, Huss RW, Thompson LC, Butz AM, Eggleston PA, Kolodner KB, Rand CS, Malveaux FJ. Moving health care education into the community. Nurs Manage. 1997 Sep;28(9):40-3. PMID 9335839
- [Background] Butz AM, Malveaux FJ, Eggleston P, Thompson L, Huss K, Kolodner K, Rand CS. Social factors associated with behavioral problems in children with asthma. Clin Pediatr (Phila). 1995 Nov;34(11):581-90. doi: 10.1177/000992289503401103. PMID 8565388